CLINICAL TRIAL: NCT06556875
Title: Regulation of HIIT Combined with IET on Vascular Function in Young Women with Normal Weight Obesity
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Beijing Sport University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: RHCIVFYWNWO
Record Dates: First submitted 2024-07-27; First posted 2024-08-16 (Actual); Last update posted 2024-10-28 (Actual); Status verified 2023-02

CONDITIONS: Normal Weight Obesity
Keywords: isometric exercise training; high-intensity interval training; normal weight obesity; vascular fitness

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- HIIT group (Active Comparator)
  Interventions: Behavioral: HIIT
- HIIT combined IET group (Active Comparator)
  Interventions: Behavioral: HIIT combined IET
- Control group (No Intervention)

INTERVENTIONS:
Behavioral: HIIT — high intensity interval training
  Arms: HIIT group
Behavioral: HIIT combined IET — high intensity interval training combined with isometric exercise training
  Arms: HIIT combined IET group

SUMMARY:
Comparison of the effects of combined IET with HIIT and HIIT on vascular function in young NWO women.

DETAILED DESCRIPTION:
This is a randomized clinical trial of single-blind with 3 arms (control group , HIIT group and IET with HIIT group), in which a pre-treatment-posttest design has been used.

ELIGIBILITY:
Inclusion Criteria:

* Female, aged between 18 and 30 years old;
* BMI between 18.5 and 24.9 kg/m2 with a BF% > 30% (normal weight obesity determination criteria);
* exercise capacity to complete the exercise programme.

Exclusion Criteria:

* Acute or chronic musculoskeletal disorders, cardiovascular diseases, etc. that prevented training;
* other diseases (such as diabetes, etc.) that had a great impact on physical condition;
* bad habits (such as smoking, drinking, etc.);
* and unstable body weight (up and down fluctuations of more than 2.5 kg) in the 3 months before the experiment.

Ages: 18 Years to 30 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 45 (Actual)
Dates: Start 2023-02-23 (Actual); Primary Completion 2023-09-30 (Actual); Study Completion 2023-12-30 (Actual)

PRIMARY OUTCOMES:
Intima-Media Thickness (IMT) | 8 weeks
  The subjects were required to sit still for 5～10 minutes before the test, and the carotid artery structural and functional parameters were recorded using a GE vivid 7 colour ultrasound instrument from the United States as follows: the subjects were required to lie in the supine position, and the probe was used to sweep longitudinally along the outer edge of the sternocleidomastoid muscle, and the maximal Intima-media thickness (IMT) was measured. Changes in Intima media thickness before and after intervention.
Flow-Mediated Dilation (FMD) | 8 weeks
  Vascular endothelial function was measured with a Japanese-made UNEX EF vascular endothelial function tester. Pressure was applied on top of the resting blood pressure and the ischaemic process was performed for 5 min. At the end of the ischaemic process, the pressure band was removed and flow-mediated dilation (FMD) of the brachial artery was calculated. Changes in Flow-mediated dilation before and after Intervention

SECONDARY OUTCOMES:
Body Composition Indicators | 8 weeks
  Body composition indicators analysis was assessed using DXA. Body composition indicators include: fat mass(kg), lean body mass(kg), percentage of body fat(%).
Body Mass Index (BMI) | 8 weeks
  Is calculated from the formula, Weight (kg) / Height2 (m2), whose unit is kg/m2. It is a rough indicator of total body fat. Changes in Body mass index before and after Intervention.
Blood Pressure (BP) | 8 weeks
  Quiet blood pressure: Systolic and diastolic blood pressures are measured using a standard mercury sphygmomanometer. Changes in blood pressure before and after intervention, including systolic blood pressure, diastolic blood pressure, and pulse pressure difference.
Pulse Wave Velocity (PWV) and ankle brachial index (ABI) | 8 weeks
  The testing instrument is Omron Atherosclerosis Tester (BP-203RPEIII). During the test, the subjects need to expose their limbs, lie flat on the bed, and keep their bodies relaxed. At the same time, they need to tie cuffs around their limbs to avoid any physical movement and ensure the accuracy of the test results. The unit of PWV is (cm/s), and ABI is a numerical value. Changes in Pulse wave velocity and ankle brachial index before and after Intervention.
Volume Oxygen Maximum (VO2max) | 8 weeks
  During the test, gradually increasing loads were performed using the Bruce running table protocol, and gas metabolism metrics were obtained at each stage of exercise using a portable Cortex-3B gas metabolism analyser. Changes in Volume oxygen maximum before and after Intervention.

CONTACTS AND LOCATIONS:
Locations (1):
- School of Sports Medicine and Rehabilitation, Beijing Sport University, Beijing, China

IPD SHARING:
Plan to Share IPD: No